CLINICAL TRIAL: NCT02768714
Title: A Randomized, Assessor-blind, Parallel Group, Multicentre Phase III Trial to Compare the Efficacy and Safety of Eurofarma's Pegfilgrastim to Neulastim® in Subjects With High Risk Stage II or Stage III / IV Breast Cancer Receiving Chemotherapy.
Brief Title: Trial to Compare the Efficacy and Safety of Pegfilgrastim Biosimilar in Subjects With High Risk Stage Breast Cancer Receiving Chemotherapy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic changes regarding the product development
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF141
Record Dates: First submitted 2016-05-09; First posted 2016-05-11 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: Breast Cancer High risk Stage II or Stage III / IV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eurofarma's pegfilgrastim (Experimental): A single 6 mg dose on Day 2 of each chemotherapy cycle of Eurofarma's pegfilgrastim (subcutaneous injection)
  Interventions: Drug: Eurofarma's pegfilgrastim
- Neulastim (Active Comparator): A single 6 mg dose on Day 2 of each chemotherapy cycle of Neulastim (subcutaneous injection)
  Interventions: Drug: Neulastim

INTERVENTIONS:
Drug: Eurofarma's pegfilgrastim — Eurofarma's pegfilgrastim is a clear, colourless solution for injection (6 mg/0.6 mL) provided in a single use prefilled syringe. Subjects randomised to Eurofarma's pegfilgrastim will receive 6 mg administered as a single SC injection in the abdomen, upper arm, or thigh on Day 2 of each CTX cycle, approximately 24 hours after
  Arms: Eurofarma's pegfilgrastim
Drug: Neulastim — Eurofarma's pegfilgrastim is a clear, colourless solution for injection (6 mg/0.6 mL) provided in a single use prefilled syringe. Subjects randomised to Eurofarma's pegfilgrastim will receive 6 mg administered as a single SC injection in the abdomen, upper arm, or thigh on Day 2 of each CTX cycle, approximately 24 hours after
  Arms: Neulastim

SUMMARY:
This is a Phase III, randomised, assessor-blind, parallel group, multicentre trial. At least 180 adult subjects with high-risk Stage II or Stage III / IV breast cancer will be randomised (1:1) to receive either Eurofarma's pegfilgrastim (n = 90) or Neulastim (n = 90) in 8 to 10 sites in Brazil. Subjects will undergo a maximum of 4 cycles of myelosuppressive chemotherapy (21 days per cycle).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Males or females ≥ 18 years of age (at the time of signing consent)
3. Breast cancer high-risk Stage II, or Stage III, or Stage IV (classification according to American Joint Committee on Cancer)
4. Eligible to receive 4 cycles of docetaxel and doxorubicin combination CTX for the treatment of high-risk stage II, III, or IV breast cancer
5. CTX-naïve
6. ECOG performance status ≤ 2
7. Adequate bone marrow function:

   * Leucocyte count < 50 x 109/L
   * ANC ≥ 1.5 x 109/L
   * Platelet count ≥ 100 x 109/L
   * Haemoglobin ≥ 10 x g/dL
8. Left Ventricular Ejection Fraction (LVEF) ≥ 50% by echocardiography or equivalent method (e.g. Multi Gated Acquisition scan) within 4 weeks prior to administration of the first dose of trial medication
9. Alanine aminotransferase and aspartate aminotransferase < 2.5 x upper limit of normal (ULN), alkaline phosphatase < 5 x ULN
10. Total bilirubin ≤ ULN
11. Creatinine ≤ 1.5 x ULN
12. Female subjects of childbearing potential must have a negative serum pregnancy test within 14 days of first dose of trial treatment and agree to use highly effective contraception (e.g. hormonal contraception or intra-uterine device [which should be established prior to the start of the trial], plus usage by at least 1 of the partners of an additional spermicide-containing barrier method of contraception) from 2 weeks prior to administration of the first dose of trial medication until trial completion, and for 30 days after the last dose of trial drug
13. Female subjects of non-childbearing potential must have a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea. A male subject with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from 2 weeks prior to administration of the first dose of trial medication until trial completion, and for 30 days after the last dose of trial drug
14. Able to comply with the trial Protocol.

Exclusion Criteria:

1. Severe chronic neutropenia
2. History of chronic myeloid leukaemia or myelodysplastic syndrome
3. History of sickle cell disease
4. Previous or concurrent malignancy except non-invasive non-melanomatous skin cancer, in situ carcinoma of the cervix, or other solid tumour treated curatively, and without evidence of recurrence for at least 10 years prior to trial entry
5. Active uncontrolled infection
6. Known human immunodeficiency virus seropositivity; active hepatitis B or hepatitis C at the Screening Visit
7. Clinically significant impairment of LVEF
8. Severe valvular heart disease, myocardial infarction, heart failure, unstable angina pectoris, uncontrolled hypertension, or uncontrolled arrhythmias within 6 months of the Screening Visit
9. Significant neurologic or psychiatric disorders including psychotic disorders, dementia, or seizures that would prohibit the understanding and giving of informed consent
10. Concurrent or prior radiotherapy within 4 weeks of the Screening Visit
11. Tumour surgery within 4 weeks prior to administration of the first dose of trial medication
12. Concurrent or prior anti-cancer treatment for breast cancer such as endocrine therapy, immunotherapy, monoclonal antibodies, and/or biological therapy
13. Concurrent prophylactic antibiotics or antibiotic treatment within 72 hours before CTX
14. Prior bone marrow or stem cell transplant
15. Previous therapy with any recombinant human granulocyte colony stimulating factor (G CSF) product
16. Known hypersensitivity to docetaxel, doxorubicin, pegfilgrastim, filgrastim, Escherichia coli proteins, or any of the excipients used in the trial medication
17. Treatment with lithium at randomization
18. Known controlled drug addiction, including alcoholism
19. Participation in a clinical trial within 30 days prior to the Screening Visit
20. Pregnant or nursing women, women planning to become pregnant, or women of childbearing potential who do not agree to use highly effective contraception (e.g. hormonal contraception or intra-uterine device [which should be established prior to the start of the trial], plus usage by at least 1 of the partners of an additional spermicide-containing barrier method of contraception) from 2 weeks prior to administration of the first dose of trial medication until trial completion and for 30 days after the last dose of trial drug
21. Male subjects with a female partner of childbearing potential who have not had a prior vasectomy and do not agree to use highly effective contraception from 2 weeks prior to administration of the first dose of trial medication until trial completion and for 30 days after the last dose of trial drug
22. Any severe concurrent disease or condition, which in the judgment of the Investigator would make the subject inappropriate for trial participation.
23. Peripheral neuropathy (sensory/motor) Grade 2 or higher (CTCAE, Version 4.03)
24. Chronic use of corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Duration of severe neutropenia (grade 4) in days during chemotherapy cycle 1. | Within the 21 Days of the first chemotherapy cycle

SECONDARY OUTCOMES:
Duration of severe neutropenia (grade 4) in days during chemotherapy Cycles 2, 3, and 4 | Four months
Incidence of febril neutropenia during chemotherapy cycles 1, 2, 3, and 4 and across all chemotherapy cycles. | Four months
Incidence of infections during chemotherapy cycles 1, 2, 3, and 4 and for all chemotherapy cycles combined. | Four months
Use of IV antibiotics to treat febril neutropenia or associated infections | Four months
Overall survival | one year after the last chemotherapy cycle